CLINICAL TRIAL: NCT01961661
Title: Effect of Probiotics on Intestinal Inflammation and Microflora in Cystic Fibrosis: a Pilot Study
Brief Title: Probiotics on Intestinal Inflammation in Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Alfredo Guarino, Full professor of Pediatrics, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CF pilot
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Cystic Fibrosis
Keywords: intestinal inflammation; intestinal microflora; children
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic (Experimental): Lactobacillus rhamnosus GG 5x10^9 colony forming units (CFU)per day
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG
- placebo (Placebo Comparator): maltodextrins
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG — Capsules containing lyophilized 6x10^9 Colony Forming Units (CFU)/die LGG, (60mg) maltodextrin (163 mg), gelatine capsule (75 mg), magnesium stearate (2 mg)
  1 capsule/die for 1 month
  Other Names: LGG
  Arms: probiotic
Dietary Supplement: placebo — Capsules containing maltodextrin (163 mg), gelatine capsule (75 mg), magnesium stearate (2 mg)
  1 cps/die for 12 months
  Arms: placebo

SUMMARY:
Cystic fibrosis (CF) is a complex systemic disease that mainly involves the respiratory and gastrointestinal (GI) tracts. The polymicrobial community composition of respiratory and GI tracts is influenced by both genetic and environmental factors. Children with CF may harbor an abnormal intestinal microflora, because of altered Cystic fibrosis transmembrane conductance regulator (CFTR) function and heavy drug load (antibiotics, pancreatic enzymes and acid suppressors). The investigators previously demonstrated that intestinal inflammation is highly frequent in CF children, being a major feature of intestinal involvement. In addition, specific probiotics significantly improved airway and GI inflammation in a preliminary trial. The aim of the study is to characterize intestinal and respiratory microflora in CF patients and to investigate the effects of daily Lactobacillus GG (LGG) supplementation on both GI and airway microflora and the eventual relationship between probiotic assumption and clinical and inflammation markers. The aim is to study the effect of microflora modification on intestinal and extraintestinal inflammation to eventually improve the quality of life of CF patients, who often suffer from intestinal and respiratory progressive disease, through a non invasive intervention consisting in the supplementation of probiotic bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF documented by sweat chloride test over 60 mmol/L and confirmed by genotype analysis with the presence of F508del/F508del or F508del/other;
* Boys and girls between 2 and 16 years of age;
* Clinical stability at enrolment, defined as no clinical evidence of acute exacerbation, no modifications in the therapeutic regimen and no hospitalization in the last 2 weeks;
* Pancreatic insufficiency;
* Basal Forced expiratory volume 1 second (FEV1) above 50% of predicted value.

Exclusion Criteria

* Colonization of respiratory tract with Burkholderia cepacia spp.;
* Steroid therapy within one month before enrolment;
* Pregnancy and fertile women taking oral contraceptives;
* Parenteral or oral antibiotics therapy within 2 weeks before enrolment;
* Regular assumption of probiotics;
* Regular assumption of azythromycin.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Modification of intestinal inflammation | baseline and after 1 month of treatment
  Evaluation of intestinal inflammation at baseline and 1 month after treatment
change in intestinal microflora composition | baseline and 1 month after treatment
  Modification of Fluorescent in Situ Hybridization profile of intestinal microflora at baseline and 1 month of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics University Federico II, Naples, Italy

REFERENCES:
- [Background] Bruzzese E, Raia V, Spagnuolo MI, Volpicelli M, De Marco G, Maiuri L, Guarino A. Effect of Lactobacillus GG supplementation on pulmonary exacerbations in patients with cystic fibrosis: a pilot study. Clin Nutr. 2007 Jun;26(3):322-8. doi: 10.1016/j.clnu.2007.01.004. Epub 2007 Mar 13. PMID 17360077
- [Background] Bruzzese E, Raia V, Gaudiello G, Polito G, Buccigrossi V, Formicola V, Guarino A. Intestinal inflammation is a frequent feature of cystic fibrosis and is reduced by probiotic administration. Aliment Pharmacol Ther. 2004 Oct 1;20(7):813-9. doi: 10.1111/j.1365-2036.2004.02174.x. PMID 15379842
- [Derived] Bruzzese E, Callegari ML, Raia V, Viscovo S, Scotto R, Ferrari S, Morelli L, Buccigrossi V, Lo Vecchio A, Ruberto E, Guarino A. Disrupted intestinal microbiota and intestinal inflammation in children with cystic fibrosis and its restoration with Lactobacillus GG: a randomised clinical trial. PLoS One. 2014 Feb 19;9(2):e87796. doi: 10.1371/journal.pone.0087796. eCollection 2014. PMID 24586292